CLINICAL TRIAL: NCT04477772
Title: A Phase I Clinical Study of Recombinant Humanized Anti-BTLA Monoclonal Antibody (JS004) in Patients With Recurrent/Refractory Malignant Lymphoma
Brief Title: A Phase I Clinical Study of JS004 in Subjects With Recurrent/Refractory Malignant Lymphoma of China
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JS004-002-I
Record Dates: First submitted 2020-07-16; First posted 2020-07-20 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Recurrent/Refractory Malignant Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Infusions, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 1mg/kg JS004, Q3W until to 2 years (Experimental): Dose escalation, enrolled 3-6 subjects
  Interventions: Biological: JS004 , Recombinant humanized IgG4k monoclonal antibody specific to BTLA for injection Intravenous infusion
- 3mg/kg JS004, Q3W until to 2 years (Experimental): Dose escalation, enrolled 3-6 subjects; Dose expansion, enrolled 9 subjects
  Interventions: Biological: JS004 , Recombinant humanized IgG4k monoclonal antibody specific to BTLA for injection Intravenous infusion
- 10mg/kg JS004, Q3W until to 2 years (Experimental): Dose escalation, enrolled 3-6 subjects
  Interventions: Biological: JS004 , Recombinant humanized IgG4k monoclonal antibody specific to BTLA for injection Intravenous infusion
- 200mg, Q3W until to 2 years (Experimental): Dose expansion, enrolled 9 subjects and indication expansion if RP2D is 200mg
  Interventions: Biological: JS004 , Recombinant humanized IgG4k monoclonal antibody specific to BTLA for injection Intravenous infusion
- 240mg JS004+100mg JS001, Q3W until to 2 years (Experimental): Dose escalation, enrolled 3-6 subjects; Dose expansion, enrolled 6-9 subjects and indication expansion if RP2D is confirmed this arm
  Interventions: Biological: JS004 , Recombinant humanized IgG4k monoclonal antibody specific to BTLA for injection Intravenous infusion; Biological: Drug：JS001, Intravenous infusion
- 240mg JS004+200mg JS001, Q3W until to 2 years (Experimental): Dose escalation, enrolled 3-6 subjects; Dose expansion, enrolled 6-9 subjects and indication expansion if RP2D is confirmed this arm
  Interventions: Biological: JS004 , Recombinant humanized IgG4k monoclonal antibody specific to BTLA for injection Intravenous infusion; Biological: Drug：JS001, Intravenous infusion

INTERVENTIONS:
Biological: JS004 , Recombinant humanized IgG4k monoclonal antibody specific to BTLA for injection Intravenous infusion — Part A: including dose escalation (1mg/kg JS004; 3mg/lg JS004; 10mg/kg JS004), dose expansion (3mg/kg JS004 and 200mg JS004) and indication expansion. Part B: including dose escalation (240mg JS004+100mg JS001; 240mg JS004+ 200mg JS001), dose expansion (240mg JS004+100mg JS001; 240mg JS004+ 200mg JS001) and indication expansion.
  Other Names: TAB004
Biological: Drug：JS001, Intravenous infusion — Part B: including dose escalation (240mg JS004+100mg JS001; 240mg JS004+ 200mg JS001), dose expansion (240mg JS004+100mg JS001; 240mg JS004+ 200mg JS001) and indication expansion.
  Arms: 240mg JS004+100mg JS001, Q3W until to 2 years; 240mg JS004+200mg JS001, Q3W until to 2 years

SUMMARY:
A First-in-human, dose-escalation, dose-expansion phase I clinical study of JS004 in subjects with recurrent/refractory malignant lymphoma in China, to evaluate the safety, tolerbility, PK, immunogenicity,antitumor activity and biomarkers of JS004, to define MTD and RP2D of JS004. A cycle is 21 days(3 weeks) which includes JS004 being administered IV Q3W and JS004 combine with JS001 being administered IV Q3W. All patients will be treated until disease progression per Lugano response critieria 2014 for Lymphoma or intolerable toxicity per CTCAE 5.0, withdrawal of consent, or end of the study, whichever occurs first. Disease progression must be confirmed at least 4 weeks but no longer than 8 weeks after initial documentation of progression.

ELIGIBILITY:
Inclusion Criteria:

1.Able to understand and sign informed consent voluntarily

2.18-70 years old

3.Pathologically confirmed malignant lymphoma

4.ECOG PS: 0-1

5.Expected survival ≥12 weeks

6.At least one measurable lesion per Lugano response critieria 2014 for Lymphoma

7.Adequate organ and marrow function, as defined below:

ANC≥1.5×109/L;

PLT≥100×109/L and ≥75×109/L for subjects with bone marrow involvement;

Hb≥90 g/L;

TBIL≤1.5 ULN, ≤2 ULN in those with hep109atic metastasis, except subjects with documented Gilbert's syndrome who must have a baseline conjugated bilirubin ≤3.0 mg/dL;

AST and ALT≤2.5 ULN, ≤5 ULN in those with hepatic metastasis;

Cr≤1.5 UL, or creatinine clearance≥50mL/min for subject;

INR ≤2 ULN and aPTT≤1.5×ULN for those with no prior anticoagulant therapy.

8.According to Fridericia's principle, QTC results need to match : Male≤450 ms，Female≤470 ms

9.Females of childbearing potential need to use effective contraception

Exclusion Criteria:

1. Patients with known allergy to macromolecular protein preparations or JS004 components
2. Prior exposure to anti-BTLA or anti-HVEM antibodies
3. Enrolled in other clinical studies within 4 weeks prior to the first dose of study treatment
4. Major surgery within 4 weeks prior to the first dose of study treatmentor still recovering from prior surgery
5. Patients who discontinued previous immunotherapy due to immune-related adverse reactions
6. Immunosuppressive agents have been used within 4 weeks prior to the first dose of study treatment
7. Prior allogeneic bone marrow transplantation or solid organ transplantation
8. Live attenuated vaccine be administered 30 days before the first dose of study treatment
9. Two or more malignancies developed within 5 years prior to first dose of study treatment
10. The patients have symptomatic, untreated, or requiring ongoing treatment central nervous system (CNS) metastases
11. Unresolved toxicities from prior anticancer therapy, defined as having not resolved to baseline or to NCI-CTCAE v5.0 Grade 0 or 1, or to levels dictated in the inclusion/exclusion criteria with the exception of alopecia.Subjects with irreversible toxicity that is not reasonably expected to be exacerbated by TAB004 may be included (e.g., hearing loss) after consultation with the medical monitor.
12. Autoimmune disease within the previous 2 years
13. A history of rapid allergic reaction, eczema, or asthma beyond the control of topical corticosteroids
14. A history of primary immunodeficiency
15. Concomitant disease that is not under control, including but not limited to: persistent or active infection, unexplained fever > 38.5°C, or heart disease, active peptic ulcer disease or gastritis
16. A history of active inflammatory bowel disease
17. HIV(+)
18. Patients with evidence of hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
19. Pregnant or lactating woman
20. Patients with vitiligo, alopecia, and hormonal replacement therapy have controlled endocrine defects
21. Any other medical factors that may affect subjects' rights, safety, compliance, ability to sign informed consent, and interpretation of study results.
22. Have a history of psychotropic drug abuse and unable to withdraw or have mental disorders.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
Number of participants and severiaty with treatment-related Adverse events as assessed by CTCAE V5.0 | 2 Years
  Safety and Tolerability

SECONDARY OUTCOMES:
Objective Response Rate (ORR) per Lugano response critieria 2014 for Lymphoma | 2 Years
Duration of Response (DOR) per Lugano response critieria 2014 for Lymphoma | 2 Years
Disease Control Rate (DCR) per Lugano response critieria 2014 for Lymphoma | 2 Years
Progrssion-free survival (PFS) per Lugano response critieria 2014 for Lymphoma | 2 Years

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China